CLINICAL TRIAL: NCT04694170
Title: Physiotherapy of Patients With Low Back Pain of Viscerovertebral Etiology.
Brief Title: Visceral Somatization and Low Back Pain.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Malá Jitka, clinical researcher of physiotherapy department, Charles University, Czech Republic
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: Sklepnikova, Kidney
Record Dates: First submitted 2020-12-26; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Lumbar Strain
Keywords: Physiotherapy; low back pain; Chinese medicine; Yoga
MeSH Terms: conditions — Sprains and Strains; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients with musculoskeletal pain in the lumbar region. Patients with typical symptoms of functional dysfunction of kidney undergo conventional physiotherapy and an alternative approach by yoga set exercising and regimen restriction according to traditional Chinese medicine.
  Interventions: Other: additional therapy; Other: conventional physiotherapy
- control group (Active Comparator): Patients with musculoskeletal pain in the lumbar region. Patients with kidney dysfunction symptoms treated by conventional physiotherapy only.
  Interventions: Other: conventional physiotherapy

INTERVENTIONS:
Other: additional therapy — Using conventional physiotherapy together with additional yoga exercising and regimen restriction acc to TCM.
  Arms: Experimental group
Other: conventional physiotherapy — Using conventional physiotherapy only.

SUMMARY:
This study aims to verify the significance of the inclusion of procedures of a comprehensive therapeutic approach according to Eastern techniques to classical physiotherapy and to find out whether these Eastern techniques can contribute to the enrichment of standard physiotherapy. According to TCM and Ayurveda, another goal is to develop appropriate regimen measures to create a yoga regimen suitable for patients who have renal and bladder dysfunction according to TCM and whose main common symptom is chronic non-specific low back pain. The study is based upon comparing a four-week physiotherapy program according to the physician's indication and a physiotherapy program enriched with compiled regimen measures and yoga exercises in selected probands.

DETAILED DESCRIPTION:
Two groups of probands were used - an experimental and control group. There were 6 probands in each group. The four-week therapy effect, which took place twice a week for 60 minutes, was compared. The control group received physiotherapy, as indicated by the physician. According to TCM and Ayurveda, the experimental group underwent physiotherapy as indicated by a doctor enriched with yoga exercises and regime measures. It was asked to perform yoga exercises daily at home. The therapy's effect was evaluated using the Short-form-36 Health-related Quality of Life Questionnaire (HRQoL), the VAS scale of pain intensity, the number of responses in the anamnestic questionnaire the author compiled the kinesiological analysis.

ELIGIBILITY:
Inclusion Criteria:

* More than half of the answers in the anamnestic questionnaire (n ≥ 14)
* More than half of the answers in the kinesiological analysis (n ≥ 7)
* Lower back pain lasting longer than 12 weeks
* Degree of pain ≥ 3 on a visual analog scale

Exclusion Criteria:

* Neurological or other structural cause of lower back or other pain key symptoms
* Serious systemic diseases (DM, heart or cancer)
* Contraindications to movements of the spine and other root joints of the body in full scope
* Pregnancy
* Simultaneous completion of another physiotherapeutic intervention, yoga exercise or treatment according to TCM
* Use of analgesics, antiphlogistics or muscle relaxants during therapy

Ages: 26 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
level of quality of life | 50 minutes
  using Short Form 36 questionnaire, minimum 100 points, less score is the sign of better quality of life, maximum = 900 points = the worst quality of life
intensity of pain | 2 minutes
  visual analog scale 0-10, 0=the best and without pain, 10=the worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Jitka Malá, PhDr.Ph.D., Principal Investigator — Charles University, Faculty of physical education and sport
Locations (1):
- Charles University, Faculty of physical education and sport, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No